CLINICAL TRIAL: NCT05177055
Title: Sleep in Psychiatric Care (SIP): A Transdiagnostic Group-based Sleep-school as Treatment for Comorbid Delayed Sleep-Wake Phase Disorder (DSWPD)
Brief Title: Sleep in Psychiatric Care (SIP): Treatment for Comorbid Delayed Sleep-Wake Phase Disorder (DSWPD)
Acronym: SIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 66304-2
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Delayed Sleep-Wake Phase Disorder; Sleep Disorder; Psychiatric Disorder
Keywords: Sleep disorders; Delayed sleep-wake phase disorder; blue-blocking glasses; psychiatric disorders; group-based treatment for circadian rhythm sleep disorder
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Sleep Wake Disorders; Mental Disorders | interventions — Waiting Lists; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Masking Description: All eligible participants will be informed that there may be a waitlist (length not specified) and receive a start-date without being informed that thay are in a waitlist group or not a waitlist group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- n=15, sleep-school 6 weeks (Experimental): Patients receive treatment as usual in the psychiatric clinic combined with participation in the sleep-school. They have already been given education on sleep regulation and sleep hygiene advice in the first meeting with the sleep-school facilitator.
  Interventions: Behavioral: Group-based light therapy at gradually advanced timing for DSWPD
- n=15, sleep-school 6 weeks and additive bb-glasses (Experimental): Patients receive treatment as usual in the psychiatric clinic combined with participation in the sleep school and additive treatment with bb-glasses. They have already been given education on sleep regulation and sleep hygiene advice in the first meeting with the sleep-school facilitator.
  Interventions: Behavioral: Group-based light therapy at gradually advanced timing for DSWPD; Behavioral: Group-based light therapy at gradually advanced timing for DSWPD and additive bb-glasses
- n=30 Six-week wait list for sleep-school (Active Comparator): Patients receive treatment as usual in the psychiatric clinic while they wait for participation in the sleep school. They have already been given education on sleep regulation and sleep hygiene advice in the first meeting with the sleep-school facilitator.
  Interventions: Other: 6-week wait list for sleep-school

INTERVENTIONS:
Behavioral: Group-based light therapy at gradually advanced timing for DSWPD — Light therapy at gradually advanced timing, Sleep education, sleep hygiene, cognitive restructuring, relaxation techniques
  Other Names: Group-LT at gradually advanced timing
  Arms: n=15, sleep-school 6 weeks; n=15, sleep-school 6 weeks and additive bb-glasses
Behavioral: Group-based light therapy at gradually advanced timing for DSWPD and additive bb-glasses — Light therapy (LT) at gradually advanced timing, bb-glasses 12 hrs after LT, Sleep education, sleep hygiene, cognitive restructuring, relaxation techniques
  Other Names: Group-LT at gradually advanced timing & bb-glasses
  Arms: n=15, sleep-school 6 weeks and additive bb-glasses
Other: 6-week wait list for sleep-school — Treatment as usual in a psychiatric outpatient clinic
  Other Names: Treatment as usual (TAU)
  Arms: n=30 Six-week wait list for sleep-school

SUMMARY:
Sleep disorders commonly co-occur with psychiatric disorders. Sleep disorders are often treated with medication or not at all in psychiatric care, although there exist a plethora of documentation of the effectiveness of sleep interventions. There is also an increase in studies showing effectiveness of sleep-interventions when the sleep disorder co-occurs with psychiatric illness. The recommended treatment for Delayed Sleep-Wake phase disorder is light therapy at gradually advanced timing and/or melatonin administered in order to help phase-advance the circadian rhythm. There is a great gap in the knowledge on how sleep disorders can be treated effectively when they occur comorbid to moderate and severe psychiatric illness. In this project the we therefore seek to investigate the effect of psychological and behavioural, group-based treatment in a randomized controlled trial (RCT) where sleep and psychiatric symptoms are the primary outcome measures.

DETAILED DESCRIPTION:
The recommended treatment for Delayed Sleep-Wake phase disorder is bright light therapy (LT) at gradually advanced timing and/or melatonin administered in order to phase-advance the circadian rhythm. Recent research has proven that dark therapy, or blocking light in wavelengths <530 nm by the use of for example orange blue-blocking glasses (bb-glasses), has shown the ability to maintain melatonin production comparable to darkness and to have an advancing effect on the circadian rhythm. The investigators therefore also want to test bb-glasses as an additive treatment to LT at gradually advanced timing.

The sleep-school at Bjørgvin District Psychiatric Hospital (DPS) is an already established treatment since 2017. The DSWPD-group gets together every other Monday from 1 pm until 3 pm. The group is open, which means that participants start at different dates and meet people in the group that might be at the end of their treatment, this often leads the group to function as a support for each other. Participants are patients at the general psychiatric outpatient clinic at Bjørgvin DPS in Bergen, Norway. Participants have been referred to the sleep-team by their psychologist or doctor. In this RCT the investigators will carry on the same structure for the group for participants that are recruited to the RCT, hence the project has high ecological validity.

All participants have an individual consultation before joining the group where the focus is on eligibility to participate in the group-based treatment, sleep-diagnostic evaluation, receive a standardized education on sleep-regulation and sleep hygiene advice and receive a date to start the group-based LT at gradually advanced timing. In a randomized manner, they will be allocated to the sleep-school group and start the treatment on the next possible date or to a 6 week wait-list and receive a date the treatment starts. All eligible participants will be informed that there may be a waitlist and receive a start-date without being informed that thay are on a waitlist group or not a waitlist group. All participants will be treated as usual (TAU) for their psychiatric problems parallel to either sleep-school or waitlist, hence both groups are in active treatment for their symptoms. Participants that start sleep-school as soon as possible, are also allocated to a) ordinary group-based LT at gradually advanced timing for 6 weeks or b) group-based group-based LT at gradually advanced timing for 6 weeks and bb-glasses. All participant will be followed up after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the sleep-school at Bjørgvin DPS psychiatric hospital
* Patients fulfilling the Diagnostic Manual for Mental Disorders (DSM-V) criteria for DSWPD comorbid to moderate to severe psychiatric illness (confirmed F-diagnosis based on the International Statistical Classification of Diseases and Related Health Problems (ICD-11) diagnostic system that are used in Norway in addition to DSWPD and/or scores of ≥19 on BDI and/or scores of ≥16 on BAI at the time of referral to the sleep school)

Exclusion Criteria:

* Night work
* Patients that do not fulfil the DSM-V criteria for DSWPD comorbid to moderate to severe psychiatric illness (confirmed F-diagnosis based on the ICD-10 diagnostic system that are used in Norway in addition to insomnia and/or scores of ≥19 on BDI and/or scores of ≥16 on BAI at the time of referral to the sleep school)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes (advancement) of sleep timing | baseline, post intervention after 6 weeks, follow-up after 12 months
  Measured by sleep diaries, Genactiv actigraphy and saliva samples (intraindividual variation of rise time (IIV), dim light melatonin onset (DLMO), rise /wake up time)

SECONDARY OUTCOMES:
Changes in objective sleep onset latency (SOL) | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by Genactive. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number of minutes of average sleep onset latency.
Changes in Sleep efficiency (SE) | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by sleep diary; total sleep time/time in bed x 100= percentage SE
Changes in Time in bed (TIB) | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by sleep diary; time from bed-time to rise time
Changes in immediate sleepiness | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by the Karolinska Sleepiness Scale (KSS). The KSS measure subjective sleepiness at a specific time point (noon). The scale gives a number from 1-9 where 9 indicates "trouble staying awake" and is the worst outcome.
Changes in objective total sleep length/time asleep (TST) | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by Genactive. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number in minutes of average total sleep time.
Work status | baseline and post intervention after 6 weeks, follow-up after 12 months
  Status of employment/unemployment, percentage disability benefits received
Changes in Total sleep length/time asleep (TST) | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by sleep diary; time in minutes from bed-time to estimated sleep onset
Changes in Early morning awakening (EMA) | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by sleep diary; minutes awake before rise time
Changes in objective sleep efficiency (SE) | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by Genactive. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number from 0-100% that gives average sleep efficiency.
Changes in objective early morning awakening (EMA) | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by Genactive. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number of average minutes early morning awakening.
Changes in well-being | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by the World Health Organisation Five Well-Being Index (WHO-5)
Changes in sleepiness | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by the Epworth Sleepiness Scale (ESS). The ESS is an 8-item scale where the respondent grades the likelihood of falling asleep or dozing off in different daily situations. The responses are graded on a 4-point likert scale 0=no likelihood to 3=very likely. A score of 11 or higher is considered an indication of excessive daytime sleepiness.
Changes in objective wake after sleep onset (WASO) | baseline and post intervention after 8 weeks, follow-up after 12 months
  Measured by Genactive. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number of average minutes awake after sleep onset.
Changes in beliefs about sleep | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by Dysfunctional Beliefs About Sleep (DBAS-16). The DBAS-16 measures the degree of dysfunctional beliefs about sleep with 16 items. It has 4 subscales (1) sleep-related worry and helplessness; 2) beliefs about sleep medications; 3) expectations about sleep need; and 4) beliefs about the consequences/effects of insomnia and 1 total scale score. The higher the score, the more dysfunctional beliefs about sleep.
Changes in Sleep onset latency (SOL) | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by sleep diary; time in minutes from bed-time to estimated sleep onset
Changes in objective time in bed (TIB) | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by Genactive. The activity recorder is worn on the wrist for 7 consecutive days. The data is downloaded to a computer program that gives the data; a number in minutes of average time in bed.
Changes in fatigue | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by the Chalders Fatigue Scale (CFS)
Changes in Sleep quality (SQ) | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by sleep diary; subjective assesment of sleep quality on a scale from 1=very light to 5=very deep
Changes in Wake after sleep onset (WASO) | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by sleep diary; minutes awake before rise time
Changes in anxiety symptoms | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by The Beck Anxiety Inventory (BAI). The BAI measure subjective symptoms of anxiety on a scale ranging from 0-63. The higher the score, the worse the anxiety.
Changes in depression symptoms | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by The Beck Depression Inventory-2 (BDI-II). The BDI measure subjective symptoms of depression on a scale ranging from 0-63. The higher the score, the worse depression.
Changes in Daytime function (DF) | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by sleep diary; subjective assesment of daytime function on a scale from 1=very good to 5=very poor
Suicide attempts and admittances in psychiatric wards | baseline and post intervention after 6 weeks, follow-up after 12 months
  Whether or not suicide has been attempted, if applicable number og attempts and whether or nor the patient has been admitted to a psychitaric ward (voluntary/forced)
Changes in anxiety and depression | baseline, bi-weekly assesment and post intervention after 6 weeks, follow-up after 12 months
  Measured by the Hospital anxiety and depression scale (HADS), Beck Depression Inventory (BDI-II) and Beck Anxiety Inventory (BAI)

OTHER OUTCOMES:
Changes in degree of experienced pain | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by a visual analogue scale (VAS Pain) ranging from 0 to 10. The higher the score, the worse the pain.
Changes in self reported emotion regulation ability | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by Difficulties in Emotion Regulation Scale (DERS) which is a 18-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores suggest greater problems with emotion regulation.
Changes in vigilance | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by the Conners Continuous Performance (CPT) Test 3rd Edition™ (Conners CPT 3™)
Changes in symptoms of inattention | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by the Adult attention deficit hyperactivity disorder (ADHD) Self-Rating Scale (ASRS). The scale contains the 18 symptoms of inattention, hyperactivity, and impulsivity defining ADHD according to the DSM-IV-TR and DSM-5. The severity of the symptoms are reported on a 5-point Likert-type scale (0-4 = never, rarely, sometimes, often, to very often), with a total range of 0-72. The higher the score, the more symptoms of inattention.
Changes in symptoms of hypochondria | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by the The Whiteley Index (WI). The 14-item WI measures assess health anxiety on a likert-scale from 1="not at all" to "5=very much". The higher the score, the more severe health anxiety.
Changes in blood pressure | baseline and post intervention after 6 weeks, follow-up after 12 months
  We will measure systolic and diastolic pressure by a digital blood pressure measurement machine.
Changes in Heart rate variability (HRV) | baseline and post intervention after 6 weeks, follow-up after 12 months
  24 -hour HRV.
Changes in work and social adjustment | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by the Work and Social Adjustment Scale (WSAS)
Changes in chronotype | baseline and post intervention after 6 weeks, follow-up after 12 months
  Measured by the Munich Chrono Type Questionnaire (MCTQ)
Client Satisfaction | post intervention after 6 weeks
  Measured by the Client Satisfaction Questionnaire (CSQ8). The CSQ-8 is an 8-item questionnaire that measures patient satisfaction with health services, where the items are rated from 1 (very low satisfaction) to 4 (very high satisfaction). The total score ranges from 8 to 32, with higher scores indicating higher degrees of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ane Wilhelmsen-Langeland, PhD, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen, Tertnes
  - Haukeland University Hospital, Bergen

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the following individual participant data (IPD); Study protocol and Informed Consent Form (ICF)
Supporting Information: Study Protocol, ICF
Time Frame: A description of when the IPD and any additional supporting information will become available and for how long, including the start and end dates or period of availability. This may be provided as an absolute date (for example, starting in January 2025) or as a date relative to the time when summary data are published or otherwise made available (for example, starting 6 months after publication).
Access Criteria: Not yet decided. PI will be reviewing requests.

REFERENCES:
- [Derived] Wilhelmsen-Langeland A, Osnes B, Gradisar M, Vagenes VA, Sorensen L, Bjorvatn B, Fasmer OB, Koenig J, Pallesen S, Saxvig IW. Group bright light therapy compared to treatment as usual for delayed sleep-wake phase disorder among patients in psychiatric care (the SIP trials): a protocol for a pragmatic, randomised controlled trial. BMJ Open. 2025 Apr 17;15(4):e093091. doi: 10.1136/bmjopen-2024-093091. PMID 40250869

DOCUMENTS (1):
  • Study Protocol (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT05177055/Prot_000.pdf